CLINICAL TRIAL: NCT00905892
Title: Metabolic Fate Modifications of Saturated Fats After an Overfeeding
Acronym: SURNUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Martine Laville PhD, MD, CRNHRA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CRNHRA-09-002
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Obesity; Lipid Metabolism; Inflammation
Keywords: overfeeding; stable isotopes; lipoprotein metabolism; lipid oxidation; fat distribution; gene expression; endotoxemia; mass spectrometry/gas chromatography
MeSH Terms: conditions — Obesity; Inflammation; Endotoxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Hyperlipidic overfeeding — 100g per day of cheese + 40g per day of almonds + 20g per day of butter

SUMMARY:
The purpose of this study is to determine the partitioning of exogenous lipids in the postprandial period while a study of overfeeding. The method is based on the incorporation of a stable isotopic tracer (d31_palmitic acid, d31_C16) in lipoprotein triglycerides (TG-CHYLOMICRON and TG-VLDL) and in free fatty acids (FFA).

DETAILED DESCRIPTION:
Healthy overweight and lean young men are subjected to an overfeeding during 56 days which corresponds to a supplement of 761 Kcal/day. During two exploration days (before : D0 et after : D56 overfeeding) they have ingested a breakfast with tracer (d31_palmitic acid, d31_C16, 20mg/kg) and blood and urine samples were collected every hour of each exploration day. The enrichment in deuterium was measured by gas chromatography-organic mass spectrometry (GC-OMS) in palmitic acid pool of lipid fractions.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years old
* BMI 18 to 30 kg/m²
* Stable physical activity
* Safety subject during medical consultation

Exclusion Criteria:

* Medical or surgical history which may affect energy expenditure (renal -cardiovascular -hepatic- endocrine-inflammatory diseases)
* Drug use that could affect energy expenditure (steroids, nicotine substitutes, thyroid hormones)
* Eating disorder
* Intensive sportive activity
* Subjects who Smoke
* Claustrophobic subjects

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Post prandial partitioning of exogenous lipids | Before and after overfeeding

SECONDARY OUTCOMES:
Genes expression in adipose and muscle tissues | Before and after overfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Martine Laville, PhD, MD, Study Director — Centre de Recherche en Nutrition Humaine Rhône-Alpes
Locations (1):
- Centre de recherche en nutrition humaine Rhone-Alpes, Pierre-Bénite, France

REFERENCES:
- [Derived] Segrestin B, Moreno-Navarrete JM, Seyssel K, Alligier M, Meugnier E, Nazare JA, Vidal H, Fernandez-Real JM, Laville M. Adipose Tissue Expansion by Overfeeding Healthy Men Alters Iron Gene Expression. J Clin Endocrinol Metab. 2019 Mar 1;104(3):688-696. doi: 10.1210/jc.2018-01169. PMID 30260393
- [Derived] Seyssel K, Alligier M, Meugnier E, Chanseaume E, Loizon E, Canto C, Disse E, Lambert-Porcheron S, Brozek J, Blond E, Rieusset J, Morio B, Laville M, Vidal H. Regulation of energy metabolism and mitochondrial function in skeletal muscle during lipid overfeeding in healthy men. J Clin Endocrinol Metab. 2014 Jul;99(7):E1254-62. doi: 10.1210/jc.2013-4379. Epub 2014 Mar 31. PMID 24684464
- [Derived] Alligier M, Meugnier E, Debard C, Lambert-Porcheron S, Chanseaume E, Sothier M, Loizon E, Hssain AA, Brozek J, Scoazec JY, Morio B, Vidal H, Laville M. Subcutaneous adipose tissue remodeling during the initial phase of weight gain induced by overfeeding in humans. J Clin Endocrinol Metab. 2012 Feb;97(2):E183-92. doi: 10.1210/jc.2011-2314. Epub 2011 Dec 7. PMID 22162470